CLINICAL TRIAL: NCT06706167
Title: Clinical Comparison Between Stainless-steel Crown, Zirconia Crown and Bioflx Crown in Primary Molars: Randomized Control Trial
Brief Title: Clinical Comparison Between Stainless-steel Crown, Zirconia Crown and Bioflx Crown in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DU0240721024
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Decayed Teeth; Carious Lesion
Keywords: primary molars; stainless steel crown; zirconia crown; bioflx crown; clinical evaluation
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: This research was designed as a randomized controlled trial conducted by a single operator to minimize operator-induced errors. A total sample of 75 primary molars was determined, allowing for potential dropouts, and was evenly distributed into three groups of 25. Each group recieved different crown, groups A for stianless steel crown, group B for zirconia crown and group C for Bioflx crown. At 6 and 12 months follow up, each crown was evaluated clinically such as plaque index , crown retentivity and gingival index.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- stainless steel crown (Active Comparator): Participants in this arm will receive stainless steel crowns for primary teeth.
  Interventions: Device: stainless steel crown; Device: Zirconia crown; Device: Bioflx crown
- zirconia crown (Experimental): Participants in this arm will receive zirconia crowns for primary teeth.
  Interventions: Device: stainless steel crown; Device: Zirconia crown; Device: Bioflx crown
- Bioflx crown (Experimental): Participants in this arm will receive Bioflex crowns for primary teeth.
  Interventions: Device: stainless steel crown; Device: Zirconia crown; Device: Bioflx crown

INTERVENTIONS:
Device: stainless steel crown — Participants in this arm received a stainless steel crown for primary teeth restoration. The crowns were selected based on the clinical assessment of the patient's dental need.
Device: Zirconia crown — Participants in this arm received a zirconia crown for primary teeth restoration. The crowns were selected to provide a more aesthetic and durable option compared to stainless steel.
Device: Bioflx crown — Participants in this arm received a Bioflx crown, which is a flexible, biocompatible material often used for pediatric crowns.

SUMMARY:
The purpose of this clinical trial was to compare clinically three different crowns for primary molars; stainless steel crown, zirconia crown and Bioflx crown.

the main questions it aims to answer are: is Bioflex crown is an alternative to stainless steel crown and zirconia crown? Seventy-five patients their age range between 3 and 8 years participated in this study. The participants are divided into three groups representing group A for stainless steel crown (n=25), group B for zirconia crown (n=25) and group C for Bioflx crown (n=25). Plaque index, crown retentivity and gingival index will be evaluated at evaluated at baseline, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient within the age group of 3-8 years old.
* Healthy children free of any systemic disease.
* Pulpotomized or pulpectomized (endodontically treated) lower second primary molars.
* Patients who have the behavioral rating of definitely positive or positive according to the frankl behaviour.

Exclusion Criteria:

* • Patient younger than 3 years old or older than 8 years old.

  * non-Healthy children or have any systemic disease.
  * primary molars with no pulpal treatment
  * Patients who have the behavioral rating of definitely negative or negative according to the frankl behaviour.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Plaque accumulation | 6 months and 12 months
  Measured using the Löe and Silness index, where each of the four surfaces of the crown (buccal, lingual, mesial, and distal) was scored from 0 to 3 (0 = no plaque, 3 = abundance of soft matter). The scores from the four areas were added and divided by four to obtain the plaque index

SECONDARY OUTCOMES:
crown retention | 6 months and 12 months
  Assessed using the USPHS criteria, where "Alpha" indicated the crown was continuous with the existing anatomic form, "Bravo" indicated a missing part of the crown but not enough to expose the underlying dentin/base, and "Charlie" indicated sufficient loss of crown substance to expose the underlying dentin/base or complete loss of the crown

OTHER OUTCOMES:
Gingival health | 6 months and 12 months
  Evaluated using the bleeding index according to Löe and Silness (1963), with scores of 0 (no inflammation), 1 (mild inflammation), 2 (moderate inflammation), and 3 (severe inflammation).

CONTACTS AND LOCATIONS:
Locations (1):
- Delta University For Science and Technology, Gamasa, El Dakhleia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
We are currently reviewing the potential for sharing individual participant data (IPD) following the completion of the study. Factors such as data privacy, participant consent, and regulatory guidelines are being considered. A final decision on data sharing will be made at the conclusion of the study, and the IPD sharing plan will be updated accordingly

REFERENCES:
- [Result] Ashima G, Sarabjot KB, Gauba K, Mittal HC. Zirconia crowns for rehabilitation of decayed primary incisors: an esthetic alternative. J Clin Pediatr Dent. 2014 Fall;39(1):18-22. doi: 10.17796/jcpd.39.1.t6725r5566u4330g. PMID 25631720
- [Result] Uhlen MM, Tseveenjav B, Wuollet E, Furuholm J, Ansteinsson V, Mulic A, Valen H. Stainless-steel crowns in children: Norwegian and Finnish dentists' knowledge, practice and challenges. BMC Oral Health. 2021 Apr 12;21(1):190. doi: 10.1186/s12903-021-01556-6. PMID 33845821
- [Result] Schuler IM, Hiller M, Roloff T, Kuhnisch J, Heinrich-Weltzien R. Clinical success of stainless steel crowns placed under general anaesthesia in primary molars: an observational follow up study. J Dent. 2014 Nov;42(11):1396-403. doi: 10.1016/j.jdent.2014.06.009. Epub 2014 Jun 30. PMID 24994618
- [Result] Seale NS, Randall R. The use of stainless steel crowns: a systematic literature review. Pediatr Dent. 2015 Mar-Apr;37(2):145-60. PMID 25905656
- [Result] Dimitrov E, Georgieva M, Andreeva RJM. Indications for use of performed crowns in pediatric dentistry. 2016;2:439-45.
- [Result] Katz CR, de Andrade Mdo R, Lira SS, Ramos Vieira EL, Heimer MV. The concepts of minimally invasive dentistry and its impact on clinical practice: a survey with a group of Brazilian professionals. Int Dent J. 2013 Apr;63(2):85-90. doi: 10.1111/idj.12018. Epub 2013 Mar 12. PMID 23550521
- [Result] Aggarwal P, Goyel V, Mathur S, Sachdev V. Effect of Stainless-Steel Crown and Preformed Zirconia Crown on the Periodontal Health of Endodontically Treated Primary Molars Correlating with IL-1beta: An In Vivo Study. J Clin Pediatr Dent. 2022 May 1;46(3):199-203. doi: 10.17796/1053-4625-46.3.5. PMID 35830632
- [Result] Kaptan A, Korkmaz E. Evaluation of success of stainless steel crowns placed using the hall technique in children with high caries risk: A randomized clinical trial. Niger J Clin Pract. 2021 Mar;24(3):425-434. doi: 10.4103/njcp.njcp_112_20. PMID 33723119
- [Result] Smail-Faugeron V, Porot A, Muller-Bolla M, Courson F. Indirect pulp capping versus pulpotomy for treating deep carious lesions approaching the pulp in primary teeth: a systematic review. Eur J Paediatr Dent. 2016 Jun;17(2):107-12. PMID 27377108
- [Result] Kopczynski K, Meyer BD. Examining Parental Treatment Decisions Within a Contemporary Pediatric Dentistry Private Practice. Patient Prefer Adherence. 2021 Mar 25;15:645-652. doi: 10.2147/PPA.S300684. eCollection 2021. PMID 33790544
- [Derived] Abdelhafez A, Dhar V. Comparative clinical performance of stainless steel, zirconia, and Bioflx crowns in primary molars: a randomized controlled trial. BMC Oral Health. 2025 Apr 18;25(1):585. doi: 10.1186/s12903-025-05869-8. PMID 40251538